CLINICAL TRIAL: NCT04200768
Title: FATLAS: Comprehensive Multi-level Characterization of Systemic and Mammary Adiposity in Breast Cancer Patients.
Acronym: FATLAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S63330
Record Dates: First submitted 2019-11-21; First posted 2019-12-16 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Body Mass Index; Adiposity; Obesity; Inflammatory Breast Cancer; Lobular Breast Cancer; Tumour Microenvironment
MeSH Terms: conditions — Breast Neoplasms; Obesity; Inflammatory Breast Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard (Other): Standard of care
  Interventions: Other: Prospective data and sample collection

INTERVENTIONS:
Other: Prospective data and sample collection — Performance of measurements of adiposity, extra collection of blood samples

SUMMARY:
FATLAS is a prospective, interventional, non Investigational Medicinal Product (IMP) study aiming to characterize the micro- and macroenvironment of breast cancer according to patient adiposity in different histological and molecular subtypes.

The macroscopic profiling of the patient's adiposity will be based on Body Mass Index (BMI), bioimpedance analysis and waist-to-hip ratio. Blood samples will be taken for lipidomic analyses and for hormonal and immuno assays. Microscopic profiling of adiposity and inflammation will be done on fresh frozen (FF) and Formalin-Fixed Paraffin-Embedded (FFPE) samples from the tumour resection specimen and will consist of histological characterization, immuno assays, multiplex immunohistochemistry, DNA sequencing and single nuclei RNA sequencing both in the tumour and in adjacent normal mammary tissue.

ELIGIBILITY:
Inclusion Criteria:

Inclusion of 30 lean (BMI 18.5 - 24.9 kg/m²), 30 overweight (BMI 25 - 29.9 kg/m²), and 30 obese (BMI ≥ 30 kg/m²) patients with histological confirmation of Invasive Ductal Carcinoma (IDC) on core diagnostic biopsy; 5 lean, 5 overweight and 5 obese Inflammatory Breast Cancer (IBC) patients; 15 lean, 15 overweight and 15 obese patients with histological confirmation of Invasive Lobular Carcinoma (ILC) on core diagnostic biopsy and 20 male subjects with any type of breast cancer that meet following criteria:

* be willing and able to provide written informed consent for this study;
* be willing to provide plasma/blood and tissue samples;
* be willing to have clinical measures of adiposity taken;
* have stage I, II or III disease (so non-metastatic) with any clinical lymph node status;
* be scheduled for surgical resection of the tumour in UZ Leuven.
* have a tumour size of ≥ 1.5 cm in order to have sufficient tumour material for the biomarker analysis. Exceptions will be made for IBC patients, as in some cases no residual tumour will be found after neoadjuvant treatment;
* be treatment naïve, i.e. not having received systemic breast cancer treatment prior to surgery. An exception is made for the IBC patients, as they will often have received first line neoadjuvant chemotherapy before surgery. IBC patients that do not undergo surgery after neoadjuvant treatment (e.g. because of inoperability of the patient) will not be included;

Exclusion Criteria:

* pregnancy at time of diagnosis;
* personal history of breast cancer (relapse/second primary);
* mixed invasive tumour type on core biopsy or special type of breast carcinoma beside pure ILC;
* history of an additional malignancy that is progressing or that has required active treatment in the 5 years prior to breast cancer diagnosis. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that have undergone potentially curative therapy or in situ cervical cancer;
* presence of an immune dysregulatory disease or condition which requires active immune modulatory treatment of any kind, or has required treatment in the past two years. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment;
* history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial in the opinion of the treating investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
BMI | Before surgery
  Calculated: body mass (kg) divided by height squared (m²)
Lipid levels in plasma | Before surgery
  Lipidomic analysis
Up- or downregulation of pathways on single cell level | At surgery
  Single nucleus RNA sequencing using 10X Genomics Platform after dissociation of tissue into single nuclei
T cell repertoire | At surgery
  Number of T-cells per population using immunohistochemical phenotypic markers of cell type and of exhaustion.
Physical activity level | Before surgery
  Time of activity of different intensities and time of sedentarity, evaluated using the Global Physical Activity Questionnaire (GPAQ) of the World Health Organisation (WHO) (scale: minutes per day, range [0 - 1440]). The higher the score for activity the better, the lower the score for sedentarity the better.
Sleep behaviour score | Before surgery
  Pittsburgh Sleep Quality Index (PSQI) score (range: [0 - 21]). Higher scores indicate worse sleep quality.
Dietary Quality Index | Before surgery
  Nutritional score (natural number, range [0 - 100]) calculated using the in-house Food Frequency Questionnaire. A score of > 70 indicates healthy dietary behaviour.
Dietary Food Intake | Before surgery
  Food intake in kcal per day calculated using the in-house Food Frequency Questionnaire.
Fat percentage | Before surgery
  Calculated from multiple frequency bio-impedance measurements (in %, range [0 - 100]).
Waist-to-hip ratio | Before surgery
  Waist circumference (cm) divided by hip circumference (cm)
Handgrip strength | Before surgery
  In kilograms (kg), measured by handheld dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No